CLINICAL TRIAL: NCT05788692
Title: "Effectiveness and Adherence to Toothbrushing Habits of Preschool Children, Using Manual or Powered Toothbrushes With or Without a Toothbrushing Assisting Application"
Brief Title: Effectiveness of Toothbrushing Habits of Preschool Children, With or Without a Toothbrushing Assisting Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Sofia Gkourtsogianni, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 523
Record Dates: First submitted 2023-03-12; First posted 2023-03-29 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Dental Plaque; Gingivitis
Keywords: plaque; toothbrush; toothbrush assisting application; children
MeSH Terms: conditions — Dental Plaque; Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: This trial is a 2x2 factorial design, since the four groups of children are formed by the cross-classification of the two factors toothbrush type (powered/manual) and use of the App (yes/no), which both have two levels.
  Children from sampled schools will be assigned randomly to one of the four experimental groups (A, B, C, D) using pre-prepared lists.
Who Masked: Investigator
Masking Description: A unique trial identification number (trial ID) will be generated for each participant, details of which will be entered into the trial management system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- electric toothbrush using a toothbrushing assisting application (Experimental): Children will be brushing with an electric toothbrush two times/day using a toothbrushing assisting application
  Interventions: Device: electric tootbrush; Device: toothbrushing assisting application
- electric toothbrush without the application (Experimental): Children will be brushing with an electric toothbrush two times/day without the toothbrushing assisting application
  Interventions: Device: electric tootbrush
- manual toothbrush using a toothbrushing assisting application (Experimental): Children will be brushing with a manual toothbrush two times /day using a toothbrushing assisting application
  Interventions: Device: manual toothbrush; Device: toothbrushing assisting application
- manual toothbrush without using the application during brushing (Experimental): Children will be brushing with a manual toothbrush two times /day without using the toothbrushing assisting application
  Interventions: Device: manual toothbrush

INTERVENTIONS:
Device: electric tootbrush — Participants will brush twice per day with an electric toothbrush
  Arms: electric toothbrush using a toothbrushing assisting application; electric toothbrush without the application
Device: manual toothbrush — Participants will brush twice per day with a manual toothbrush
  Arms: manual toothbrush using a toothbrushing assisting application; manual toothbrush without using the application during brushing
Device: toothbrushing assisting application — Participants will brush twice per day with toothbrushing assisting application
  Arms: electric toothbrush using a toothbrushing assisting application; manual toothbrush using a toothbrushing assisting application

SUMMARY:
The aim of this study is to investigate the effectiveness of the use of a toothbrushing assisting mobile application in dental plaque removal and adherence to the toothbrushing routine, in preschool children (3-5 yrs old) when brushing with either manual or powered toothbrush.

Objectives: To identify the effectiveness in dental plaque control in relation to the following parental characteristics:

* Sociodemographic (area of residence, average income, education level)
* Oral Health status
* Oral Health Literacy
* Parenting style
* Parental oral hygiene practices

DETAILED DESCRIPTION:
This is a single blind randomized clinical trial with 6 months follow up that involves:

1. Written parental informed consent for their child's participation in the study
2. Completion of self-administered parental questionnaires on: (i) medical and dental history of the child, demographics, parental attitudes and oral hygiene practices, and child's diet and oral hygiene practices and (ii) Parenting style, using Parenting Styles Dimensions Questionnaire (PSDQ)
3. Completion, by face-to-face interview, of the Oral Health Literacy instrument (GROHL) validated for Greek language.
4. Oral hygiene and toothbrushing instructions to both parents and children
5. Toothbrushing at home using manual or powered toothbrushes with and without the use of a toothbrushing assisting app.
6. Dental examination of the children regarding oral hygiene status (plaque), gingivitis and dental caries, pre and post the intervention period.

Sample: Parent-child dyads will be recruited from pre-schools in areas of various socio-economic status of Attica. To avoid recruiting the same parent twice, only one child from each family will be recruited as long as the child fulfils the above criteria

Procedures -Informed Consent and Questionnaires:

Prior to the school examination date, written consent forms and questionnaires will be sent to the parents of all groups and will be returned to the school completed in order for the children to take part in the examination.

A) Questionnaire on socioeconomic characteristics (e.g. region of origin, education level, financial status), demographic characteristics (age, gender), medical history and medication received, dental history (regarding previous dental examination and treatment, oral hygiene, and diet habits), parental attitudes and oral hygiene practices as well as oral health status of the parent. The questionnaire has been previously used and validated in Greek.

B) The Parenting Styles Dimensions Questionnaire (PSDQ) is a validated tool to evaluate the parenting styles of children aged 4-12 years and has been widely used in various populations. The tool consists of 32 statements assessing parental reactions to child behaviour. The authoritarian domain is measured by 12 statements, the authoritative domain by 15 statements and the permissive domain by 5 statements. Parents rank each statement on a 5-point Likert scale as to how often they exhibit each behavior. The PSDQ has been translated and validated in Greek.

Dental education: Children of all groups meeting eligibility criteria for the study will receive oral hygiene instructions, such as toothbrushing twice-daily (day and night) with a fluoride toothpaste (pea-sized amount, 1000ppmF-) for two minutes and healthy eating habits.

Dental examination: Clinical examination of soft and hard oral tissues will be performed by an experienced paediatric dentist and will be completed in the classrooms with artificial light using a mouth mirror and a periodontal probe. Findings will be recorded in standardized form. Patient's data will be coded with a number in order to maintain blinding and confidentiality (personal details, age, sex and the study group). Before examination all children will receive information regarding the examination in a playful way and become familiar with the dental instruments and the procedure.

The following will be recorded:

Dental plaque accumulation, Calculus, Gingivitis and Dental Caries

Calibration for dental plaque assessment will be done using 20 photographs of teeth stained following application of a two-tone disclosing solution. Photographs will be assessed by the examiner prior to study initiation and after a two week interval to determine intra-reliability. The examiner will be calibrated for dental caries as well. Intra-observer repeatability will be tested as the examiner will repeat clinical examination at a 2 two week interval in 20 numbers of patients routinely treated in the postgraduate clinic of Paediatric Dentistry for their dental needs.

Allocation to groups : Children from particular schools will be selected randomly on individual basis. Each subject will brush for 6 months as follows:

Group A: electric toothbrush using a toothbrushing assisting application Group B: electric toothbrush without the application Group C: a manual toothbrush using a toothbrushing assisting application Group D: a manual toothbrush without using the application during brushing

The sample of children will be stratified by gender and caries status (presence of cavitated lesions). There will thus be 2 x 2 = 4 strata each with a corresponding random list of group assignments (for example, D A B C C A D B D C A B ….). For every eligible child that enters the study we first check to which stratum they belong. Then the investigators will apply to that child the next unused group assignment in the corresponding list. For example, using the list above, the first child of that stratum to enter the study goes into experimental group D, the next into group A, the next into group B, and so on. As each list consists of repeated random permutations of the set of four groups A, B, C, and D, each of these groups will appear with approximately equal frequency in each stratum.

Oral hygiene instructions to parents : Parents will be given detailed brushing instructions depending on the type of toothbrush they are using (electric brush /manual) to brush their child's teeth and the use of the app. This will be done in a one-to-one meeting between a designated dentist and the parent using an online communication platform. In this session the Greek-language OHL instrument (GROHL) - translated and validated in Greek -will also be completed by interview. Furthermore parent's questions regarding oral health issues will be addressed.

In addition, parents will be able to get prevention advice for their children by contacting an assigned oral health care professional of the department via email or telephone contact.

Follow up examinations:

One month: In this examination the following parameters will be recorded: dental plaque, calculus, gingivitis. The examination will be done without prior brushing or cleaning of the teeth.

6 months: In this examination the following parameters will be recorded: dental plaque, calculus, gingivitis. The examination will be done without prior brushing or cleaning of the teeth. A questionnaire about brushing and any adverse effects or problems they had from the procedure will be completed. Furthermore, questions on the importance of professional guidance on the use of power brushes (trough the electronic platform) and the improved brushing behaviour within the parents will be included.

Data collection will be carried out in the kindergarten under standard dental epidemiological conditions. All data will be collected on paper using specific report forms and identified solely by each subjects' trial ID. Then data will be saved in electronic forms on secure University servers with access limited to study investigators. The paper consent forms and paper record sheets will be held separately and securely in a controlled access area in locked cabinets.

Sample size : sample required for the study was calculated using the G*Power 3 program (version 3.1.9.4). The calculation was carried out for the case of testing effects in a 2-way ANOVA, for example, for the examination of a quantitative outcome such as Plaque Index in relation to the combination of toothbrush type (powered or manual) and use of the App (yes or no). Conventional values were used for the input parameters, namely, significance level α = 0.05, power = 1 - β = 0.80 and effect size = 0.25 (medium). The required total sample size for this configuration was 128 subjects, that is, 32 children in each of the 4 groups. With a slightly bigger effect size (0.3), the sample size could be reduced to 90 (22-23 per group). An additional 2-3 extra children per group would allow for potential losses to follow up. Therefore, the recommended target sample size is preferably 35 children per group (total 140), with a minimum of 25 (total 100).

Statistical analysis : This trial is a 2x2 factorial design, since the four groups of children are formed by the cross-classification of the two factors toothbrush type (powered/manual) and use of the App (yes/no), which both have two levels. A principal method of analysis will therefore be 2-way ANOVA carried out on the plaque score and other quantitative outcome variables, or on their changes from baseline. Within this framework, it is possible to investigate simultaneously the effect of toothbrush type, the effect of using the App, and their interaction - that is, whether the size of the effect of toothbrush type depends on whether or not the App is used. The sample size calculations in this proposal have been carried out for F tests in these ANOVAs.

In addition, regression analyses or ANCOVA will be carried out for the relation of outcome variables to items recorded at baseline, including scale scores obtained from the questionnaires completed by the parents.

Ethical considerations: Verbal and written information will be given to children (appropriate for their age) and their parents in all groups and parental Informed Consent will be obtained. Parents/caregivers will have the opportunity to state that they do not want their child to participate. The forms will be returned to school in a closed envelope to ensure that unauthorized persons cannot see the completed forms.

All information collected will be kept strictly confidential and process of all personal data (i.e. socio-demographic characteristics, medical & dental history, and questionnaire responses) will comply with all aspects of the General Data Protection Regulation (GDPR). A unique trial identification number (trial ID) will be generated for each participant, details of which will be entered into the trial management system.

Adverse events: Due to the nature of participant involvement, no serious adverse events are anticipated that will be related to the trial. However, the following procedures will be undertaken to capture any complications associated with the trial. Parents will be informed in the participant information sheet that they are able to report any concerns or anything out of the ordinary that has happened to them as a result of taking part in the trial, to the research team during the course of the study. Contact details of the main researcher will be provided. All children will get an explanation in a playful way and become familiar with the dental instruments and examination process.

Details of any serious adverse events or adverse events reported by the participants will be considered by the principal investigators and research team.

ELIGIBILITY:
Inclusion Criteria:

* children 3-5 years of age
* good general health
* born in Greece and understand Greek language
* at least 16 fully erupted primary teeth with facial and lingual surfaces that can be scored (erupting teeth will not be scored).
* living in the same household with the parent consenting for participation in the study

Exclusion Criteria:

* any medical condition or medications that affect gingival condition (e.g. antiepileptics)
* tooth surfaces that plaque cannot be scored due to extensive carious lesions
* presence of abscess or fistula , pain or need for urgent dental treatment
* difficulties in communication due to language issues
* lack of cooperation
* use of powered toothbrush in the past

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline of mean Plaque score in one month | one month
  According to TURESKY QUIGLEY/HEIN plaque index: '0' = No plaque present, '1' = Separate flecks of plaque at the cervical margin, '2' = A thin continuous band of plaque (up to 1 mm) at the cervical margin,'3'= A band of plaque wider than 1 mm but covering less than one-third of the side of the crown of the tooth. '4' = Plaque covering at least one-third but less than two-thirds of the side of crown of the tooth, '5' = Plaque covering two-thirds or more of the side of the crown of the tooth.
Change from baseline of Gingival Index score in one month | one month
  Gingivitis according to Gingival Index (GI) by Löe - Silness, on 6 sites of teeth.Scoring criteria for GI are 0=Normal gingival, 1=Mild inflammation slight change in color, slight edema, no bleeding on probing, 2=Moderate inflammation, redness, edema and glazing, bleeding on probing, 3=Severe inflammation, marked redness and edema, ulceration, tendency for spontaneous bleeding.
Change from baseline of Calculus Index score in one month | one month
  Will be recorded using Calculus Surface Index (CSI). Presence (=0) or absence (=1) of calculus on the lingual surface of the lower 4 anterior teeth will be assessed by visual examination with mouth mirror and the percentage of the surfaces with calculus to those examined in total will be recorded for each individual
Change in times of brushing in one month | one month
  Will be collected via a checklist
Change from baseline of mean Plaque score in six months | six months
  According to TURESKY QUIGLEY/HEIN plaque index: '0' = No plaque present, '1' = Separate flecks of plaque at the cervical margin, '2' = A thin continuous band of plaque (up to 1 mm) at the cervical margin,'3'= A band of plaque wider than 1 mm but covering less than one-third of the side of the crown of the tooth. '4' = Plaque covering at least one-third but less than two-thirds of the side of crown of the tooth, '5' = Plaque covering two-thirds or more of the side of the crown of the tooth.
Change from baseline of Gingival Index score in six months | six months
  Gingivitis according to Gingival Index (GI) by Löe - Silness, on 6 sites of teeth.Scoring criteria for GI are 0=Normal gingival, 1=Mild inflammation slight change in color, slight edema, no bleeding on probing, 2=Moderate inflammation, redness, edema and glazing, bleeding on probing, 3=Severe inflammation, marked redness and edema, ulceration, tendency for spontaneous bleeding.
Change from baseline of Calculus Index score in six months | six months
  Will be recorded using Calculus Surface Index (CSI). Presence (=0) or absence (=1) of calculus on the lingual surface of the lower 4 anterior teeth will be assessed by visual examination with mouth mirror and the percentage of the surfaces with calculus to those examined in total will be recorded for each individual
Change in times of brushing in six month | six months
  Will be collected via a checklist

SECONDARY OUTCOMES:
Change from baseline in mean dmft score in 6 months | six months
  Dental caries will be based on the ICDAS II criteria (International Caries Detection and Assessment System), converted subsequently to dmft/DMFT -the highest ICDAS score will be used for the conversion to dmft. The D/d component of the dmft index will be broken down into two subcomponents, incipient lesions (ICDAS 1-2) and progressed lesions (ICDAS 3-6). Missing teeth will be scored only if they are extracted due to caries. Restorations will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sotiria Gizani, Study Chair — Associate Professor and Head, Department of Paediatric Dentistry, School of Dentistry, NKUA; William Papaioanou, Study Director — Associate Professor, Department of Preventive and Community Dentistry, School of Dentistry, NKUA; Andreas Agouropoulos, Study Director — Assistant Professor, Department of Paediatric Dentistry, School of Dentistry, NKUA
Locations (6):
- Greece (6):
  - Paidikos Stathmos of 251 Air Force General Hospital, Athens
  - A Paidikos Stathmos NKUA, Athens
  - B Paidikos Stathmos NKUA, Athens
  - 3rd Paidikos Stathmos Vrilissia, Vrilissia
  - 4th Paidikos Stathmos Vrilissia, Vrilissia
  - 1st Paidikos Stathmos Vrilissia, Vrilissia

IPD SHARING:
Plan to Share IPD: No